CLINICAL TRIAL: NCT06468787
Title: ECHO-009 Kosmos Anatomical Object Labeling and View Identification Pivotal Study
Brief Title: Kosmos Anatomical Object Labeling and View Identification Pivotal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EchoNous Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECHO-009
Record Dates: First submitted 2024-06-06; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Disorder; Hepatic Disorder; Spleen Disorder; Kidney Disorder; Pulmonary Disorder; Renal Disorder; Hepatobiliary Disorders; GYN Disorders
MeSH Terms: conditions — Heart Diseases; Digestive System Diseases; Splenic Diseases; Kidney Diseases; Lung Diseases; Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Anatomical Object Labeling and View Identification Comparison (Experimental): Labeling and identification comparative assessment
  Interventions: Device: Kosmos Anatomical Object Labeling and View Identification Algorithms

INTERVENTIONS:
Device: Kosmos Anatomical Object Labeling and View Identification Algorithms — Participants underwent limited ultrasound scanning by both cardiac sonographers and abdominal sonographers. Algorithm's performance on the view identification task and the object labeling task is compared to majority opinion of 5 radiologists.

SUMMARY:
This is a multi-site, multi-group study that obtained two sets of ultrasound scans from all enrolled participants. Participants underwent limited ultrasound scanning by both cardiac sonographers and abdominal sonographers. Algorithm's performance on the view identification task and the object labeling task is computed.

ELIGIBILITY:
Inclusion Criteria:

* Persons able to:
* Read and sign an English consent form.
* Give consent for participation.
* Able and willing to comply with study requirements.
* Those aged 18 years through 89 years, healthy as well as individuals with pathology, including but not limited to:
* Persons with heart-related conditions such as myocardial or pericardial disease.
* Persons with lung-related conditions such as: asthma, COPD, bronchitis, pulmonary fibrosis, sarcoidosis, pulmonary hypertension, pulmonary hypertension, bronchiectasis, lung cancer, pneumonia, pulmonary edema, pulmonary embolism
* Persons with abdomen-related conditions such as: pancreatitis, gastroesophageal reflux disease, irritable bowel syndrome, colitis, gastroenteritis, ulcers, abdominal aortic aneurysm, splenomegaly, liver disease, kidney disease.

Exclusion Criteria:

* Children (minors) under 18 years old
* Adults over 89 years old
* Pregnant individuals
* Those who cannot or refuse to sign their consent
* Those who cannot provide informed consent
* Those who cannot speak or read English
* Vulnerable populations, i.e., individuals whose willingness to participate in the study could be unduly influenced by the expectation of medical benefits associated with participation
* Individuals with mobility issues that prevent them from having an echo examination
* Individuals with severe chest deformities, or other critical clinical situations, e.g., life critical urgent situations where there is no time for anything else than what is needed for patient care, that prevent them from having an echo examination.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
False discovery rate of the anatomical object labeling function on expert-obtained images | Post data acquisition (3 months)
  The objective of this study is to compare the average frame-level disagreement of object labeling by majority opinion of five expert reviewers. The frame-level disagreement is defined as False Discovery Rate as in (1) FDR = 1-Precision=FP/(FP+TP) (1) Where TP≡True Positive and FP≡False Positive. A True Positive is counted when the majority opinion of five expert reviewers agrees with the location of predicted labels in the image. A False Positive counted when majority opinion of five expert reviewers disagrees with the location of one or more predicted labels.
  False Discovery Rate (FDR) is measured for a particular image frame between predicted objects and the majority opinion of five reviewers. The frame-level FDR threshold for this prospective study is 20%. Therefore, for a successful outcome the frame-level FDR must be less than 20%.
False discovery rate of the anatomical view identification function on expert-obtained images | Post data acquisition (3 months)
  The objective of this study is to compare the average frame-level disagreement of object labeling by majority opinion of five expert reviewers. The frame-level disagreement is defined as False Discovery Rate as in (1) FDR = 1-Precision=FP/(FP+TP) (1) Where TP≡True Positive and FP≡False Positive. A True Positive is counted when the majority opinion of five expert reviewers agrees with the location of predicted labels in the image. A False Positive counted when majority opinion of five expert reviewers disagrees with the location of one or more predicted labels.
  False Discovery Rate (FDR) is measured for a particular image frame between predicted objects and the majority opinion of five reviewers. The frame-level FDR threshold for this prospective study is 20%. Therefore, for a successful outcome the frame-level FDR must be less than 20%.

CONTACTS AND LOCATIONS:
Overall Officials: Asad Karim, MD, Principal Investigator — Revival Research Institute LLC
Locations (1):
- REVIVAL research institute, LLC, Sherman, Texas, United States